CLINICAL TRIAL: NCT02730130
Title: A Multicenter Single Arm Phase II Study to Assess the Efficacy of Pembrolizumab Plus Radiotherapy in Metastatic Triple Negative Breast Cancer Patients
Brief Title: Study to Assess the Efficacy of Pembrolizumab Plus Radiotherapy in Metastatic Triple Negative Breast Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Cedars-Sinai Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-032
Record Dates: First submitted 2016-03-29; First posted 2016-04-06 (Estimated); Results first posted 2019-10-04 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer; Metastatic Triple Negative
Keywords: Pembrolizumab; Radiotherapy; 16-032
MeSH Terms: conditions — Breast Neoplasms | interventions — pembrolizumab; Radiotherapy

ARMS (1):
- Pembrolizumab Plus Radiotherapy (Experimental): Subjects will receive pembrolizumab 200 mg as an IV infusion. RT begins D1 prior to dose 1 of Pembrolizumab. Pembrolizumab will be administered as a 30 minute IV infusion. Radiotherapy will be performed using external beam ionizing radiation as standard therapy in accordance with institutional standard practice. The dose of radiation will be a standard regimen/fractionation used in palliation: 3000 cGy, delivered in five 600 cGy fractions within 5-7 days.
  Interventions: Drug: Pembrolizumab; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Pembrolizumab
Radiation: Radiotherapy

SUMMARY:
The purpose of this study is to find out what effects, good and/or bad, pembrolizumab has on the patient and areas of cancer in their body that did not receive radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent/assent for the trial.
* Be female ≥ 18 years of age on day of signing informed consent.
* Histologically or cytologically-confirmed TNBC (defined as ER <1%, PR <1%, her-2-neu 0-1+ by IHC or FISH-negative or as per MD discretion) at each enrolling institution.
* Metastatic or locally recurrent TNBC.
* Subjects who are resistant to conventional chemotherapy or have declined conventional therapy for TNBC. Patients having received any prior line of systemic therapy for inoperable/recurrent or metastatic disease are eligible.
* At least one tumor for which palliative RT is considered appropriate standard therapy.
* At least one index lesion that will not undergo RT and which is measurable based on RECIST 1.1.
* If an archived tumor tissue is available, be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1 of RT.
* Repeat palliative RT will be permitted for the treatment of isolated, non-target lesions.
* Consent for blood draws for research purposes.
* Consent for use of available archived tissue for research purposes.
* Have a performance status of 0 or 1 on the ECOG Performance Scale.
* Demonstrate adequate organ function; all screening labs should be performed within 28 days (+7 days) of treatment initiation, unless otherwise indicated.

Hematological

* Absolute neutrophil count (ANC) ≥1.5, k/mcL
* Platelets ≥100 k,/ mcL
* Hemoglobin ≥9 g/dL or ≥5.6 mmol/L without transfusion or EPO dependency (within 7 days of assessment) Renal
* Serum creatinine OR Measured or calculated^a creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 X upper limit of normal (ULN) OR ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN Hepatic
* Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
* AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases
* Albumin ≥2.5 mg/dL Coagulation
* International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants ≤1.5 X ULN unless subject is receiving anticoagulant therapy
* Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants
* Female subject of childbearing potential should have a negative pregnancy test or documentation of absence of pregnancy by a gynecologist within 2 weeks of initiating radiation therapy.
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.

Note: ^aCreatinine clearance should be calculated per institutional standard.

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has a known history of active TB (Bacillus Tuberculosis)
* Hypersensitivity to pembrolizumab or any of its excipients.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≥ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy or targeted small molecule therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≥ Grade 1 or at baseline) from adverse events due to a previously administered agent.

Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.

* If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Has a known additional malignancy that progressed or required treatment in the last 5 years. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain parenchymal metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis, which is excluded regardless of clinical stability.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has known history of/active, non-infectious pneumonitis requiring treatment with steroids or has history of/active interstitial lung disease.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or has participated in another Merck pembrolizumab clinical trial.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days of planned start of study therapy.

Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-06-03 (Actual); Primary Completion 2017-09-26 (Actual); Study Completion 2022-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Barker, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Memorial Sloan Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering at Mercy Medical Center, Rockville Centre, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Pembrolizumab Plus Radiotherapy: Subjects will receive pembrolizumab 200 mg as an IV infusion. RT begins D1 prior to dose 1 of Pembrolizumab. Pembrolizumab will be administered as a 30 minute IV infusion. Radiotherapy will be performed using external beam ionizing radiation as standard therapy in accordance with institutional standard practice. The dose of radiation will be a standard regimen/fractionation used in palliation: 3000 cGy, delivered in five 600 cGy fractions within 5-7 days.
  Pembrolizumab
  Radiotherapy
Period: Overall Study
Arm/Group | Pembrolizumab Plus Radiotherapy
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab Plus Radiotherapy
Number analyzed (Participants) | 17
Age, Continuous [Median (Full Range); unit: years] | 52 [37 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 12
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate in Unirradiated Lesions
Description: RECIST v. 1.1 criteria will be used.
Time Frame: 13 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab Plus Radiotherapy
Number analyzed (Participants) | 17
Participants
  Complete Response | 3
  Partial Response | 0
  Stable Disease | 1
  Progressive Disease | 8
  Not Evaluable | 5

2. Secondary Outcome: Duration of Response
Description: Only participants with a Complete Response and a Partial Response will be evaluated.
Time Frame: 13 weeks
Measure: Median (Full Range); unit: months
Arm/Group | Pembrolizumab Plus Radiotherapy
Number analyzed (Participants) | 3
months | 4.5 [4.1 to 8.3]

3. Secondary Outcome: Time to Response
Description: Only participants with a Complete Response and a Partial Response will be evaluated.
Time Frame: 13 weeks
Measure: Median (Full Range); unit: months
Arm/Group | Pembrolizumab Plus Radiotherapy
Number analyzed (Participants) | 3
months | 2.8 [2.7 to 3.0]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Pembrolizumab Plus Radiotherapy
All-Cause Mortality (participants affected / at risk) | 15/17
Serious Adverse Events (participants affected / at risk) | 17/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab Plus Radiotherapy (N=17)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Fatigue (General disorders) | 5
Alanine aminotransferase increased (Investigations) | 1
Thromboembolic event (Vascular disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Platelet Count Decreased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Fever (General disorders) | 2
Insomnia (Psychiatric disorders) | 1
Soft tissue infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab Plus Radiotherapy (N=17)
Infection (Infections and infestations) | 1
Lymphopenia (Investigations) | 2
Biliary obstruction (Hepatobiliary disorders) | 1
Bilirubinemia (Investigations) | 1
Radiation Dermatitis (Injury, poisoning and procedural complications) | 1
Fatigue (General disorders) | 2
Skin Changes (Skin and subcutaneous tissue disorders) | 2
Nausea (Gastrointestinal disorders) | 2
ALT increased (Investigations) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Localized edema (General disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-11): https://cdn.clinicaltrials.gov/large-docs/30/NCT02730130/Prot_SAP_000.pdf